CLINICAL TRIAL: NCT04479878
Title: Observational and Monocentric Study of Complications in Adults With Cancer Receiving an Artificial Parenteral Nutrition in the Central Vein Initiated in Hospitalization
Brief Title: Complications in Adults With Cancer Receiving an Artificial Parenteral Nutrition in the Central Vein
Acronym: ONAC
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: ICM2013/40
Record Dates: First submitted 2020-07-06; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Cancer
Keywords: parenteral nutrition
MeSH Terms: conditions — Neoplasms; Hyperphagia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will evaluate the frequency of complications in adult cancer patients with central venous parenteral nutrition and the identification of aggravating factors.

DETAILED DESCRIPTION:
In oncology, central venous catheters are used for treatments such as chemotherapy, hydration, antibiotic therapy and parenteral nutrition. However, these catheters are responsible for serious complications often infectious or vascular. They can lead to suspension or discontinuation of treatments and can lead to life-threatening outcomes for patients. The incidence rate and risk factors for central venous catheter-related infections in oncology remain poorly known. Recently, a prospective study targeted a 5-fold increase in the risk of catheter infection when parenteral nutrition was associated with chemotherapy.

This is why the indications of parenteral nutrition must be respected and enteral nutrition promoted where possible.

the investigator conducted a retrospective study in 1998 over 10 years and 6 months, including all patients who received or received a parenteral nutrition at home, for at least one month.

Of 153 patients with implantable sites, 181 infectious episodes were recorded in 68 patients (44.4% of the population) with an estimated median infection rate of 2 infections/patients (1-12). There was a clear predominance of community-borne skin germs (85% Staphylococcus sp and 3% multi-resistant bacteria (BMR)).

In order to improve our nursing practices, and reduce complications for patients,the investigator propose the establishment of an observatory of complications in adults with cancer benefiting from superior parenteral nutrition on the central venous tract initiated in hospitalization with a planned return home

ELIGIBILITY:
Inclusion Criteria:

* Central venous parenteral nutrition initiated in hospitalization with a planned return home (with parenteral nutrition).
* Life expectancy > 3 months
* OMS (World Health Organization) performance status (PS) 0, 1 or 2
* With initial dietary consultation during hospitalization
* Age ≥ 18 years
* Hospitalized 48 hours or more
* Patient Information and Signature of Informed Consent
* patient must be affiliated to a French Social Security System

Exclusion Criteria:

* OMS> 3 or 4
* Patient in the process of infection
* Patient followed up in surgery
* Patient without central vein
* Patient with superior cave thrombosis,
* Inability to undergo medical follow-up of the trial for geographical, social or psychological reasons,
* Terminally ill palliative patient, excluding surgery.
* Patient whose regular follow-up is not possible due to psychological, family, social or geographical reasons; • Medical or psychological condition which, in the opinion of the investigator, will not allow the patient to complete the study or sign informed consent with full knowledge (Article L.1121-6, L.1121-7, L. 1211-8, L. 1211-9);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient With Cancer Receiving an Artificial Parenteral Nutrition in the Central Vein
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Prospective assessment of infectious and vascular complications in parenteral nutrition on implanted venous device through systematic registration in relation to care practices | from date of inclusion visit until an average of 1 year
  Number and date of infectious complications per patient
Prospective assessment of infectious and vascular complications in parenteral nutrition on implanted venous device through systematic registration in relation to care practices | from date of inclusion visit until an average of 1 year
  Number and date of vascular complications per patient

SECONDARY OUTCOMES:
Assessment of care practices | from date of inclusion visit until an average of 1 year
  Assessment of Nurse's Handwashing Every Two Weeks (10-point note)
Assessment of care practices | from date of inclusion visit until an average of 1 year
  Evaluation of the consumption of sterile sets (for connections and disconnections on the Central Venous Way) and Huber needles by the provider every two weeks (note on 10 points)
Assessment of care practices | from date of inclusion visit until an average of 1 year
  Evaluation of pulsed rinse after nutrition by the nursing office - question asked only once at the end of observation ("never" - "sometimes to often" - "always")
Evaluation of hospitalizations and central vein ablations | from date of inclusion visit until an average of 1 year
  Collection of the number of hospitalizations
Evaluation of hospitalizations and central vein ablations | from date of inclusion visit until an average of 1 year
  Collection of the duration of hospitalizations
Evaluation of compliance with protocols for the medical care of infectious and vascular complications | from date of inclusion visit until an average of 1 year
  assessment of adherence to protocols for the management of infectious and vascular complications on a 5-point scale corresponding to the 5 main recommended international steps for infectious complications, and on 1 point (yes/no) according to the parenteral nutrition treaty for vascular complications
Evaluation of serious complications related to the central vein | from date of inclusion visit until an average of 1 year
  number of complications related to the central vein per patient

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lacroix, Study Chair — ICM Val d'Aurelle
Locations (1):
- Icm Val D'Aurelle, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toure A, Vanhems P, Lombard-Bohas C, Cassier P, Pere-Verge D, Souquet JC, Ecochard R, Chambrier C. Totally implantable central venous access port infections in patients with digestive cancer: incidence and risk factors. Am J Infect Control. 2012 Dec;40(10):935-9. doi: 10.1016/j.ajic.2012.01.024. Epub 2012 May 26. PMID 22633131
- [Result] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Result] O'Grady NP, Alexander M, Dellinger EP, Gerberding JL, Heard SO, Maki DG, Masur H, McCormick RD, Mermel LA, Pearson ML, Raad II, Randolph A, Weinstein RA. Guidelines for the prevention of intravascular catheter-related infections. The Hospital Infection Control Practices Advisory Committee, Center for Disease Control and Prevention, U.S. Pediatrics. 2002 Nov;110(5):e51. doi: 10.1542/peds.110.5.e51. PMID 12415057
- [Result] Ullmann AJ, Cornely OA, Donnelly JP, Akova M, Arendrup MC, Arikan-Akdagli S, Bassetti M, Bille J, Calandra T, Castagnola E, Garbino J, Groll AH, Herbrecht R, Hope WW, Jensen HE, Kullberg BJ, Lass-Florl C, Lortholary O, Meersseman W, Petrikkos G, Richardson MD, Roilides E, Verweij PE, Viscoli C, Cuenca-Estrella M; ESCMID Fungal Infection Study Group. ESCMID* guideline for the diagnosis and management of Candida diseases 2012: developing European guidelines in clinical microbiology and infectious diseases. Clin Microbiol Infect. 2012 Dec;18 Suppl 7:1-8. doi: 10.1111/1469-0691.12037. PMID 23137133